CLINICAL TRIAL: NCT01341743
Title: A Multi-center, Randomized, Controlled Study to Evaluate the Efficacy and Safety of Generic Entecavir Monotherapy or in Combination With Adefovir for Chronic Hepatitis B Patients With Inadequate Response to NUC Therapy
Brief Title: Efficacy Optimizing Research of Chronic Hepatitis B Patients With Inadequate Response to NUC Therapy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: JiangSu Chia-Tai Tianqin Pharmacy Co.Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MOH-04
Record Dates: First submitted 2011-02-16; First posted 2011-04-26 (Estimated); Last update posted 2013-10-30 (Estimated); Status verified 2013-09

CONDITIONS: Hepatitis B
Keywords: chronic hepatitis B; inadequate response; NUC therapy
MeSH Terms: conditions — Hepatitis B; Hepatitis B, Chronic | interventions — entecavir; adefovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A (Active Comparator): oral entecavir 1mg daily for 104 weeks
  Interventions: Drug: Entecavir
- B (Active Comparator): oral entecavir 1mg daily and adefovir 10mg daily for 104 weeks
  Interventions: Drug: Entecavir, Adefovir
- C (Active Comparator): oral entecavir 0.5mg daily and adefovir 10mg daily for 104 weeks
  Interventions: Drug: Entecavir, Adefovir

INTERVENTIONS:
Drug: Entecavir — patients will receive oral entecavir 1mg, daily for 104 weeks.
  Arms: A
Drug: Entecavir, Adefovir — patients in this arm will receive oral entecavir 1mg daily and adefovir 10mg daily for 104 weeks
  Arms: B
Drug: Entecavir, Adefovir — patients in this arm will receive oral entecavir 0.5mg daily and adefovir 10mg daily for 104 weeks
  Arms: C

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of generic entecavir monotherapy or in combination with adefovir for chronic hepatitis B patients with inadequate response to NUC therapy

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18-65 years;
* Capable of understanding and signing the informed consent. Willing to comply with the study requirements;
* Serum HBsAg positive and ALT<10ULN at study screening;
* Patients have been treated with one nucleoside/nucleotide analogue for more than 6 months and are still on treatment;

Exclusion Criteria:

* History of viral breakthrough or genotypic resistance on previous therapy;
* History of decompensated liver function, or current signs/symptoms of decompensation e.g. ascites, variceal bleeding, encephalopathy or spontaneous peritonitis;
* Patient has a history of hepatocellular carcinoma(HCC) or findings suggestive of possible HCC;
* Other protocol defined exclusion criteria.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2010-12; Primary Completion 2014-06 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
proportion of subjects with hepatitis B virus (HBV)DNA<300copies/ml at week 104 | week 104

SECONDARY OUTCOMES:
serum HBV DNA reduction from baseline at week 104 | week 104
The proportion of subjects with ALT normalization at week 104 | week104
The proportion of subjects with HBeAg loss and seroconversion at week 104 | week104
The proportion of subject with HBsAg loss and seroconversion at week 104 | week104
The proportion of subjects with mutations of rtN236T/A181V, rtL180M/rtM204V/rtT184/rtS202 and/or rtM250 at week 104 | week104

CONTACTS AND LOCATIONS:
Overall Officials: JinLin Hou, MD, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (16):
- China (16):
  - Beijing Ditan Hospita, Beijing, Beijing Municipality
  - Beijing Friendship Hospital Attached to the Capital Medical University, Beijing, Beijing Municipality
  - Department of infectious disease, First Hospital of Peking University, Beijing, Beijing Municipality
  - People'S Hospital Under Beijnig University, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - The First People's Hospital of Foshan, Foshan, Guangdong
  - Department of infectious disease, Nanfang Hospital, Guangzhou, Guangdong
  - GuangDong Provincial People's hospital, Guangzhou, Guangdong
  - First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Tongji Hospital of Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Xiangya Hospital Central-South Univrsity, Changsha, Hunan
  - First Hospital .Jilin Unniversity, Changchun, Jilin
  - ShengJing Hospital of China Medical University, Shenyang, Liaoning
  - Changhai Hospital affiliated to Second Military Medical University, Shanghai, Shanghai Municipality
  - Huashan Hospital，Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Ruijin Hospital, Shanghai, Shanghai Municipality